CLINICAL TRIAL: NCT00211536
Title: A Randomized, Active Control, Multi-Center Study Comparing the Effect of Intraperitoneal Insulin Administration to Subcutaneous Insulin Administration on Glycemic Control and the Frequency of Severe Hypoglycemia
Brief Title: Study Comparing Effectiveness of Intraperitoneal Insulin Administration to Subcutaneous Insulin Administration
Acronym: MIP310
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Medtronic Diabetes (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CE-025A6
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Results first posted 2011-06-23 (Estimated); Last update posted 2011-09-21 (Estimated); Status verified 2011-08

CONDITIONS: Type 1 Diabetes
Keywords: Diabetes; Implantable Insulin Pump; Intraperitoneal Insulin Delivery
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MiniMed Implantable insulin Pump (MIP) (Experimental): The experimental group will receive intraperitoneally (IP) delivered insulin via the Medtronic MiniMed Implantable Pump (MIP). At the time of implant, the pump will be filled with Aventis HOE21PH U400 insulin and the subject will be treated with this insulin for the first 180 days post implant. During the refill procedure performed 180 days post implant, any insulin remaining in the pump will be removed and the pump will be refilled with Medtronic MiniMed Implantable Pump Human Recombinant Insulin.
  Interventions: Drug: Medtronic MiniMed Implantable Pump Human Recombinant Insulin; Device: Medtronic MiniMed Implantable Pump System; Drug: Aventis HOE21PH U400
- Subcutaneous insulin arm (SC) (No Intervention): The control group will remain on their current pre-study subcutaneous insulin therapy of either Multiple Daily Injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII - external insulin pump). The SC group will not be restricted to the type of insulin used, or be required to change or modify their current diabetes therapy for the purpose of the study.

INTERVENTIONS:
Drug: Medtronic MiniMed Implantable Pump Human Recombinant Insulin — 400 IU per ml - dosage based on the Investigators clinical judgement and the individual subject requirements.
  Other Names: Human insulin injection (rDNA origin)
  Arms: MiniMed Implantable insulin Pump (MIP)
Device: Medtronic MiniMed Implantable Pump System — The implantable pump system is intended to provide continuous intraperitoneal delivery of insulin in subjects with diabetes.
  Other Names: IP insulin pump system
  Arms: MiniMed Implantable insulin Pump (MIP)
Drug: Aventis HOE21PH U400 — 400 IU per ml - dosage based on the Investigators clinical judgement and the individual subject requirements.
  Other Names: Aventis U400 insulin; Aventis ETP Insulin
  Arms: MiniMed Implantable insulin Pump (MIP)

SUMMARY:
The purpose of this study is to evaluate the effectiveness of insulin delivered in the peritoneum (abdomen)by an implantable pump in Type 1 diabetics.

DETAILED DESCRIPTION:
Implantable insulin delivery pumps have been shown to reduce the occurrence of severe hypoglycemia in Type 1 DM subjects, as demonstrated in numerous European studies. Glycemic control is difficult to attain in subjects using exogenous insulin due to the risk of severe hypoglycemia. This study is aimed at comparing the efficacy of intraperitoneal (IP) insulin therapy to intensive subcutaneous insulin therapy over a period of 12 months.

ELIGIBILITY:
* Type 1 diabetes mellitus (American Diabetes Association definition)
* HbA1c greater than or equal to 7.5%
* Intensive insulin treatment for at least 3 months
* Physical and intellectual ability to operate MIP system
* Subject has been under the routine care of the investigator for at least two months prior to enrollment
* Subject has a reliable support person (defined as a person who has daily contact with the subject and knows whom to contact in the event of an emergency).
* Capability and willingness to perform self-monitoring of blood glucose at least four times daily for 9 months of the study and 7 times daily for 3 months of the study
* Physical and intellectual ability to operate the MIP system and to comply with the data reporting requirements of the study.
* Subject is willing to sign the informed consent form (approved by local Institutional Review Board and Medtronic MiniMed)

Exclusion Criteria:

* The subject's insulin usage exceeds 66 units per day.
* Severe complications such as advanced autonomic neuropathy, legal blindness, or symptomatic cardiovascular disease as evidenced by a cardiovascular episode within the last six months
* Reside at or plan to travel to elevations above 8000 feet during the study period (commercial airline travel is acceptable)
* Subject who is pregnant, of childbearing potential or lactating and is neither surgically sterile, using contraceptives (devices, oral or implanted) nor other physician approved contraceptive
* The subject has any major concomitant disease or any physical or psychological disorder within the last five years, which might be considered life threatening, or which might confound the collection or interpretation of the study data
* The subject has previously enrolled in or participated in an investigational drug or device study within the preceding 4 weeks
* The subject has any condition that precludes him/her from completing the study requirements
* Has plans for activities which require them to go 25 feet below sea level

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2002-06; Primary Completion 2004-08 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Lee, MD, Study Director — Medtronic
Locations (5):
- United States (5):
  - Sansum Medical Research Institute, Santa Barbara, California
  - University of Colorado Health Sciences Center, Aurora, Colorado
  - Hellman & Rosen Endocrine Associates, North Kansas City, Missouri
  - Cleveland Clinic, Wooser, Ohio
  - Diabetes & Glandular Disease Clinic, San Antonio, Texas

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Centers were either university or clinic based endocrinology centers. The centers were required to recruit from their current patient population. This ensured that they had knowledge of the medical and behavioural history prior to enrollment. The experimental pumps were to be implanted and so the study could not be blinded.
Pre-assignment Details: All subjects trained on testing for Low Blood Glucose Index (LBGI) and a baseline collection of this data for all subjects was collected prior to a block randomization plan. The randomization visit occured 14 days prior to the study start, to allow for scheduling of the implantation surgery for those randomized to the MIP arm.
Groups:
- MiniMed Implantable Insulin Pump (MIP): The experimental group will receive intraperitoneally (IP) delivered insulin via the Medtronic MiniMed Implantable Pump (MIP). At the time of implant, the pump will be filled with Aventis HOE21PH U400 insulin and the subject will be treated with this insulin for the first 180 days post implant. During the refill procedure performed 180 days post implant, any insulin remaining in the pump will be removed and the pump will be refilled with Medtronic MiniMed Implantable Pump Human Recombinant Insulin.
  The primary efficacy analysis set will include all subjects randomized and followed, at least, to Visit 5 (90 days, first insulin refill for MIP group). Missing data are treated as missing. There is no extrapolation or interpolation of missing values. This set is considered to be the As-Treated Data Analysis Set and is the primary data set used in the analysis.
- Subcutaneous Insulin Arm (SC): The control group will remain on their pre-study subcutaneous insulin therapy either Multiple Daily Injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII - external insulin pump). The SC group will not be restricted to the type of insulin used.
  For consistency, results were analyzed for subjects that completed beyond V5. These were considered to be the "As Treated" group.
  The primary efficacy analysis set will include all subjects randomized and followed, at least, to Visit 5 (90 days, first insulin refill for MIP group). Missing data are treated as missing. There is no extrapolation or interpolation of missing values. This set is considered to be the As-Treated Data Analysis Set and is the primary data set used in the analysis.
Period: Overall Study
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC)
Started | 53 | 54
As Treated Data Analysis Set | 52 (This set includes all subjects followed to Visit 5 (90 days, first insulin refill for MIP group).) | 48
Completed | 49 | 47 (This set includes all subjects followed to Visit 5 (90 days, first insulin refill for MIP group).)
Not Completed | 4 | 7
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Physician Decision | 0 | 5
Not completed — Adverse Event | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC) | Total
Number analyzed (Participants) | 52 | 48 | 100
Age, Categorical [Count of Participants; unit: Participants] — This set includes all subjects followed to Visit 5 (90 days, first insulin refill for MIP group).
  Participants
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 52 | 48 | 100
    >=65 years | 0 | 0 | 0
Age Continuous [Mean (Standard Deviation); unit: years] — Results reported on the As-Treated Data Analysis set (n=100). This is the primary efficacy analysis set and will include all subjects randomized and followed, at least, to Visit 5. Missing data are treated as missing. There is no extrapolation or interpolation of missing values.
  years | 43.3 (10.8) | 40.7 (11.9) | 42 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31 | 31 | 62
  Male | 21 | 17 | 38
Region of Enrollment [Number; unit: participants]
  United States | 52 | 48 | 100

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c and Compared Between Groups
Description: To determine whether Intra Peritoneal insulin delivery via MIP results in glycemic control that is equal to or superior (i.e. not inferior to) control with SC therapy (Ho : μ (IP) -μ (SC) ≥ 0.50% A1C), a repeated measures analysis of variance, adjusting for baseline A1C using SAS Proc Mixed was used to compare average A1C trends over time between the two treatment groups (19). Type 3 Least Square (LS) means for each group were assessed. The Estimate statement within SAS proc mixed was used to estimate contrasts among the LS means and confidence intervals for the contrasts.
Time Frame: Baseline and 12 months
Population: The primary efficacy analysis set is the As treated data set and includes all subjects randomized and followed, at least, to Visit 5 (90 days, first insulin refill for MIP group). Missing data are treated as missing. There is no extrapolation or interpolation of missing values.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC)
Number analyzed (Participants) | 52 | 48
percent HbA1c | -0.3122449 (0.8908406) | 0.1191489 (0.8691921)
Statistical Analysis 1: Comparison: MiniMed Implantable Insulin Pump (MIP) vs Subcutaneous Insulin Arm (SC); Sample size calculations were performed on the primary endpoint: the average glycosylated hemoglobin (A1C). Sample size was estimated using a two-sample, one-sided t-test with a significance level of 0.05. The projected sample size of 50 subjects per treatment group provides 79% power to reject the null hypothesis in favor of the alternative hypothesis that the average A1C in both the MIP and SC groups are equivalent, assuming an effect size of 0.50% and a standard deviation of 1.0%; Test type: Non-Inferiority or Equivalence — For the average A1C, the goal was to show non-inferiority of MIP compared to SC. The minimal clinically relevant increase in A1C (%) was set at 0.50%. The between-subjects standard deviation of A1C was assumed to be 1.0% based on previous studies; p < 0.05, Mixed Models Analysis; Repeated measures analysis of variance, adjusting for baseline A1C using SAS Proc Mixed to compare A1C trends over time between the treatment groups; Least square means = 0.3, 95% CI 1-sided [upper limit 0.5], Standard Error of Mean 0.2

2. Primary Outcome: Incidence of Severe Hypoglycemia Events
Description: The total number of severe hypoglycemia events, defined as a clinical episode of hypoglycemia (resulting in seizure or coma, requiring hospitalization, intravenous glucose or glucagon administration), or any hypoglycemia that requires assistance from another person, compared between the two study arms from Baseline to 12 months.
Time Frame: 12 months
Population: The primary efficacy analysis set will include all subjects randomized and followed, at least, to Visit 5 (90 days, first insulin refill for MIP group). Missing data are treated as missing. There is no extrapolation or interpolation of missing values. This set is considered to be the As-Treated Data Analysis Set for the purpose of analysis.
Measure: Number; unit: events
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC)
Number analyzed (Participants) | 52 | 48
events | 2 | 4

3. Secondary Outcome: Average Daily Blood Glucose
Description: For each subject, a minimum of two blood glucose readings per day was required for calculation of the average daily mean. The overall mean of the mean for each subject for the measure time frame was then calculated. The mean of the results for all subjects in each group were then analyzed and compared between groups both at Baseline and 12 months.
Time Frame: average from baseline to 12 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC)
Number analyzed (Participants) | 52 | 48
mg/dL | 186.77 [182.7 to 190.83] | 195.8 [192.01 to 199.58]

4. Secondary Outcome: Mean Amplitude of Glycemic Excursions (MAGE)
Description: MAGE was calculated by taking the arithmetic mean of BG excursions when both ascending and descending segments of the curve exceed one Standard Deviation of the average 24-hour BG value. MAGE was calculated for each subject using SMBG data from periods in which subjects had a minimum of 4 and maximum of 10 readings daily. The overall mean of the mean for each subject for the measure time frame was then calculated. The mean of the results for all subjects in each group were then analyzed and compared between groups both at Baseline and 12 months.
Time Frame: average from baseline to 12 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC)
Number analyzed (Participants) | 52 | 48
mg/dL | 136.27 [131.07 to 141.47] | 149.2 [143.09 to 155.31]

5. Secondary Outcome: Low Blood Glucose Index (LBGI);
Description: 4 to 10 daily blood glucose readings (BG) were required for this measure. LBGI was calculated from BG values collected for 30 days prior to Visit 2 and 30 days following Visits 5 and 7. The continuous measure was compared between the two treatment groups for the three periods with a repeated measures ANOVA using proc mixed. Type 3 least square means for each group were assessed and estimate statements used to make comparisons among the LS means and create confidence intervals on the contrasts.
Time Frame: average from baseline to 12 months
Population: as for outcome 2
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC)
Number analyzed (Participants) | 52 | 48
mg/dL | 2.14 [1.85 to 2.44] | 2.27 [1.94 to 2.61]

ADVERSE EVENTS:
Time Frame: Adverse event data collected from screening at 30 days prior to randomization until end of study phase at one year.
Groups:
- MiniMed Implantable Insulin Pump (MIP): The experimental group will receive intraperitoneally (IP) delivered insulin via the Medtronic MiniMed Implantable Pump (MIP). At the time of implant, the pump will be filled with Aventis HOE21PH U400 insulin and the subject will be treated with this insulin for the first 180 days post implant. During the refill procedure performed 180 days post implant, any insulin remaining in the pump will be removed and the pump will be refilled with Medtronic MiniMed Implantable Pump Human Recombinant Insulin.
  Results were analyzed for subjects that completed beyond V5, which was the end of the first 90 day period of IP insulin therapy. These were considered to be the "As Treated" group.
  All randomized subjects were assessed for safety risk.
- Subcutaneous Insulin Arm (SC): The control group will remain on their pre-study subcutaneous insulin therapy either Multiple Daily Injections (MDI) or Continuous Subcutaneous Insulin Infusion (CSII - external insulin pump). The SC group will not be restricted to the type of insulin used.
  For consistency, results were analyzed for subjects that completed beyond V5. These were considered to be the "As Treated" group. All randomized subjects were assessed for safety risk.
Arm/Group | MiniMed Implantable Insulin Pump (MIP) | Subcutaneous Insulin Arm (SC)
Serious Adverse Events (participants affected / at risk) | 9/53 | 7/54
Other Adverse Events (participants affected / at risk) | 51/53 | 27/54
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiniMed Implantable Insulin Pump (MIP) (N=53) | Subcutaneous Insulin Arm (SC) (N=54)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Central Line Infection (Infections and infestations) | 1 (1) | 0 (0)
Diabetes Mellitus aggravated (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Diabetes out of control
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 2 (2) | 2 (4)
Multiple Myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Operation NOS (Surgical and medical procedures) | 3 (3) | 0 (0) — Pump explanted for unknown reason
Post procedual site infection (Surgical and medical procedures) | 1 (1) | 0 (0)
Road traffic Accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skin ulcer (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2.5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MiniMed Implantable Insulin Pump (MIP) (N=53) | Subcutaneous Insulin Arm (SC) (N=54)
Hyperglycemia NOS (Metabolism and nutrition disorders) | 11 (13) | 4 (4)
Hypoglycemia NOS (Metabolism and nutrition disorders) | 13 (23) | 1 (2)
Nasopharygitis (Infections and infestations) | 9 (12) | 6 (8)
Seasonal allergy (Immune system disorders) | 5 (8) | 2 (2)
Upper respiratory tract infection NOS (Infections and infestations) | 11 (14) | 8 (9)
Urinary tract infection (Renal and urinary disorders) | 5 (5) | 6 (7)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days